CLINICAL TRIAL: NCT06750978
Title: Feasibility and Effects of Behavioral Interventions to Reduce Problematic Smartphone Use (PSU) with College Students
Brief Title: Interventions for PSU Among College Students
Acronym: PSU
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Wen Anthony, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2024000027; AWD00012208 (Other Grant/Funding Number: Rutgers Research Council)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Problematic Smartphone Use
Keywords: Problematic smartphone use, smartphone overuse

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with repeated measures design will be used. The study consists of three phases. (1) Baseline phase (2 weeks): Following eligibility screening and consent, all participants will install an app developed by the research team. The app will track and report participants daily smartphone usage and establish a baseline pattern of PSU. (2) Experimental phase (4 weeks): After the baseline data collection, participants will be randomized on a rolling basis into one of the four conditions (12 participants in each condition): Self-Reflection, Self-Reflection + Alternative Activity Engagement, Self-Reflection + Contingency Management, and Control. Participants daily smartphone usage, review of usage data, and/or evidence of alternative activity engagement will be recorded by the app and reported to the researcher. (3) Follow-up phase (2 weeks): The three intervention conditions will be withdrawn in this phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Self-reflection (Experimental): Participants actively review their smartphone usage data each day, which will be verified by the app.
  Interventions: Behavioral: Self-reflection
- Self-reflection + Alternative activity engagement (Experimental): Participants actively review their smartphone usage and engage in alternative activities which are identified by the participants, which will be recorded and verified via the app.
  Interventions: Behavioral: Self-reflection + Alternative activity engagement
- Self-reflection + Contingency management (Experimental): Participants will actively review their smartphone usage each day, which will be verified via the app. If the participant meets their daily PSU reduction goal, they will receive an incentive ($8); if they do not meet their goal, they will receive nothing.
  Interventions: Behavioral: Self-reflection + Contingency management
- Control (No Intervention): Participants will not engage in any behavioral intervention strategies

INTERVENTIONS:
Behavioral: Self-reflection — Participants will be guided to identify goals of daily PSU reduction. o Participants will be guided to actively review their smartphone usage data each day.
  Arms: Self-reflection
Behavioral: Self-reflection + Alternative activity engagement — Participants will be guided to identify goals of daily PSU reduction and actively review their smartphone usage data each day. Participants will be guided to develop a plan for alternative activity engagement and confirm their engagement in the alternative activities as planned.
  Arms: Self-reflection + Alternative activity engagement
Behavioral: Self-reflection + Contingency management — Participants will be guided to identify goals of daily PSU reduction and actively review their smartphone usage data each day. Participants will receive an incentive ($8) if they meet the daily PSU reduction goal.
  Arms: Self-reflection + Contingency management

SUMMARY:
This project proposes to evaluate the feasibility and effects of behavioral intervention strategies on problematic smartphone use among college students. The project proposes to evaluate three behavioral intervention components- self-reflection via actively monitoring phone usage, increasing engagement in non-smartphone activities, and contingency management (i.e., financial incentives) - on short-term and long-term reductions in problematic smartphone use (PSU) among college students.

The research team will develop a mobile application, referred to as the app, to collect data on a subject's daily phone usage and activity engagement. The app will comprise three features, with specific sets of features being activated during different phases.

* Feature 1: The app will autonomously track the time spent on the apps categorized as social media and gaming.
* Feature 2: The app will display the daily amount of usage on social media and gaming apps, with an option for a subject to confirm their acknowledgment of the daily time spent.
* Feature 3: The app will display an option for subject to confirm their engagement in the alternative activities as planned.

DETAILED DESCRIPTION:
This project will extend previous research by investigating whether alternative activity engagement and contingency management in combination with self-reflection via actively monitoring smartphone usage produce greater reductions in PSU, compared to self-reflection alone. Further, this study aims to compare the feasibility and effects of two low-cost behavioral intervention components (i.e., self-reflection and increasing alternative activity engagement) to those of a high-cost intervention component (i.e., contingency management) among university students.

Research questions:

1. What are the effects of self-reflection, alternative activity engagement, and contingency management in reducing the severity of problematic smartphone use?
2. What is the feasibility and acceptability of the various intervention strategies?

Research hypothesis:

1. Participants who receive the self-reflection intervention will have a greater reduction in their PSU compared to participants who receive no intervention.
2. Participants who receive the intervention combining self-reflection and alternative activity engagement will have a greater reduction in their PSU compared to participants who receive no intervention and participants who receive only self-reflection intervention.
3. Participants who receive the intervention combining self-reflection and contingency management will have a greater reduction in their PSU compared to participants who receive no intervention and participants who receive only self-reflection intervention.

College students who are 18+ years old, use an Android smartphone, identified as having problematic smartphone use (scored 31+ on the Smartphone Addiction Scale), and interested in learning strategies to reduce unwanted smartphone use are eligible for participation.

Intake session: Research subjects who are eligible for participation will meet with a designated graduate student research assistant for consent and app installation. Subjects who provide consent and meet the eligibility criteria will be asked to install the app that will be used to track a subject's daily smartphone usage and their engagement in assigned interventions. The intake meeting will be about 10-30 minutes. Following the consent and eligibility screen, subjects will also be randomly assigned to one of the four conditions, including three intervention conditions and one control condition. The randomization will be conducted by the PI.

2-week baseline phase: Following the intake session, subjects' daily smartphone usage will be tracked for two weeks to establish baseline data. During this phase, only Feature 1 of the app will be activated.

4-week intervention phase: After the 2-week baseline phase, subjects who are assigned to intervention conditions will meet with the designated graduate student research assistant to learn about the intervention strategy, identify goals of daily PSU reduction, and update the app for an assigned condition. This meeting will be about 30 minutes to 1 hour.

* Subjects who are assigned to Condition 1(Self-reflection) will be guided to actively review their smartphone usage data each day. In this condition, Features 1 and 2 of the app will be activated.
* Subjects who are assigned to Condition 2 (Self-reflection + Alternative activity engagement) will be guided to develop a plan for alternative activity engagement. Each day, subjects will actively review their smartphone usage and engage in alternative activities as planned. In this condition, Features 1, 2, and 3 of the app will be activated.
* Subjects who are assigned to Condition 3 (Self-reflection + Contingency management) will be guided to actively review their smartphone usage data each day. If the subject meets their daily PSU reduction goal, they will receive an incentive ($8) that day; if they do not meet their goal, they will receive nothing. In this condition, Features 1 and 2 of the app will be activated.
* Subjects who are assigned to Condition 4 (Control condition) do not engage in any active intervention. Their daily smartphone usage will be tracked using the app. In this condition, only Feature 1 of the app will be activated.

At the end of the 4-week intervention phase, subjects will be asked to complete an online survey that assesses their severity of PSU. Subjects who receive interventions will also be asked about their involvement, acceptability, and satisfaction with the assigned intervention.

2-week follow-up phase: After the 4-week intervention phase, subjects will be asked to stop the assigned intervention. Subjects' daily smartphone usage will be tracked for additional 2-weeks to establish follow-up data. In this condition, only Feature 1 of the app will be activated.

ELIGIBILITY:
Inclusion Criteria:

* Rutgers students who are 18+ years old
* Use an Android smartphone
* identified as having problematic smartphone use (scored 31+ on the Smartphone Addiction Scale)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Daily smartphone usage data | 8 weeks
  The amount of time spent on apps identified by the participants
Problematic smartphone use | 8 weeks
  Severity of problematic smartphone use will be assessed with the Smartphone Addiction Scale (SAS) short version. The SAS short version includes 10 items. The sum of these items gives an overall score ranging 10-60, with higher score indicating more severe problematic smartphone use.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Anthony, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns about maintaining participant privacy and confidentiality. Although measures such as data anonymization can reduce re-identification risks, complete elimination of such risks cannot be guaranteed. Additionally, the consent forms used in this study do not include provisions for IPD sharing. To comply with ethical guidelines and regulatory standards, we have decided not to share IPD at this time.